CLINICAL TRIAL: NCT03908307
Title: A 12-month, Open-label, Multicenter, Phase 4 Study to Evaluate the Efficacy and Safety of OZURDEX® Implant 700 µg (Dexamethasone) on Patients With Macular Edema Secondary to Retinal Vein Occlusion in China (YANGTZE Study)
Brief Title: Evaluation of OZURDEX® in Patients With Macular Edema Secondary to Retinal Vein Occlusion in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMO-MA-EYE-0575
Record Dates: First submitted 2019-03-28; First posted 2019-04-09 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Eye (Experimental): OZURDEX implant 700 μg
  Interventions: Drug: OZURDEX

INTERVENTIONS:
Drug: OZURDEX — Implant 700 μg

SUMMARY:
This study will take place in China to evaluate the safety and efficacy of OZURDEX implant 700 μg in the treatment of macular edema due to retinal vein occlusion (RVO) in patients who have never received treatment for RVO.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Patient diagnosed with macular edema due to RVO (either BRVO or CRVO, non-ischemic)
* Retinal thickness ≥ 300 μm by SD-OCT in the central 1 mm macular subfield of the study eye at the Screening visit
* BCVA score of 19 to 73 letters (approximately 20/400 to 20/40 Snellen equivalent) in the study eye measured by ETDRS method at Screening
* < 3 months of macular edema duration
* Treatment-naive patients (ie, have not previously received any treatment for macular edema secondary to RVO)

Exclusion Criteria:

* Uncontrolled systemic disease
* Presence of/history of any ocular condition other than macular edema that affects visual acuity (eg, cataract, severe macular ischemia, foveal atrophy, age-related macular degeneration, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass syndrome, prior macular detachment)
* Any of the following ≤ 3 months before study entry or anticipated need within the coming 3 months:
* Intraocular surgery
* Laser photocoagulation
* Intraocular injection
* Periocular steroid injection
* Vitrectomized eye
* Aphakic eyes with ruptured posterior lens capsule or presence of an ACIOL, iris or transscleral fixated intraocular lens
* History of marked IOP elevation in response to steroid treatment that (a) required IOP-lowering treatment, (b) resulted in a >10 mm Hg increase in IOP from predose, or (c) resulted in IOP >25 mm Hg
* History of glaucoma or ocular hypertension (IOP > 21 mm Hg), or optic nerve head change consistent with glaucoma damage, and/or glaucomatous visual field loss in the study eye (patients with a history of previous angle closure that has been successfully treated with either a laser or surgical peripheral iridotomy [PI] are allowed as long as the visual fields have been stable for > 1 year prior to study entry and the patient has been and can be safely dilated).
* Any active ocular infection (i.e., bacterial, viral, parasitic, or fungal) in either eye at the Screening visit
* Female patients who are pregnant, nursing, or planning a pregnancy, or who are of childbearing potential and not using a reliable means of contraception
* Any condition that may interfere or preclude participation in the study
* Use of systemic steroids (e.g., oral, intravenous, intramuscular, epidural, rectal, or extensive dermal) within 1 month prior to Baseline or anticipated use at any time during the study (inhaled, intranasal, and intra-articular/intrabursal corticosteroids are allowed)
* Use of immunosuppressants, immunomodulators, antimetabolites, and/or alkylating agents within 3 months prior to Baseline or anticipated use at any time during the study
* Use of warfarin or heparin within 2 weeks prior to Baseline or anticipated use within the study period
* Known allergy, hypersensitivity or contraindication to the study medication, its components, fluorescein or povidone iodine
* Current enrollment in another drug or device study within 30 days prior to Baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-09-26 (Actual); Study Completion 2021-09-26 (Actual)

PRIMARY OUTCOMES:
Mean change in visual acuity from Baseline | At Month 6
  Determined by best corrected visual acuity (BCVA)
Proportion of patients with a BCVA improvement of 15 letters or more compared to Baseline | At Month 6
  Measured using the ETDRS visual acuity protocol
BCVA average change from Baseline in area under the curve (AUC) analysis | At Month 6

SECONDARY OUTCOMES:
Mean change from Baseline in BCVA | After first follow-up visit, at each injection, and at Month 12
Mean change from Baseline in Central Retinal Thickness (CRT) | At Months 6 and 12
Mean change from Baseline in the National Eye Institute (NEI) Visual Function Questionnaire (VFQ)-25 | At Months 6 and 12
  25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better functioning. Original numeric values from the survey will be recoded with the worst and best possible scores set at 0 and 100 points, respectively. In this format, scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score.
Mean number of OZURDEX injections | During the 12-month study
Mean retreatment interval in months | During the 12-month study
Proportion of patients with 2nd injection | During the 12-month study
Proportion of patients with 3rd injection | During the 12-month study
Time to 2nd injection | During the 12-month study
Time to 3rd injection | During the 12-month study
Correlation between the change of BCVA and extent of leak by fluorescein angiography (FA) | At Month 6

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (9):
- China (9):
  - Peking Union Medical College Hospital /ID# 233616, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, CMU /ID# 233608, Beijing
  - The First Xiangya Hospital of Central South University /ID# 233627, Changsha Hunan
  - The First Affiliated Hospital of Dalian Medical University /ID# 233688, Dalian
  - Qilu Hospital of Shandong University /ID# 233605, Jinan
  - The Eye and ENT Hospital Affiliated of Fudan Univesity /ID# 233666, Shanghai
  - Shanghai General Hospital /ID# 233579, Shanghai
  - Joint Shantou International Eye Center of Shantou University and The Chinese Uni /ID# 233580, Shantou
  - Tianjin Eye Hospital /ID# 233581, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=CMO-MA-EYE-0575&Latitude=&Longitude=&LocationName=#additional-resources-section